CLINICAL TRIAL: NCT05481281
Title: Comparison Of Dexmedetomidine And Ketamine For Control Of Shivering In Vaginal Hysterectomy Proceeded Under Spinal Anesthesia
Brief Title: Comparison Of Dexmedetomidine & Ketamine For Control Of Shivering In Vaginal Hysterectomy Under Spinal Anesthesia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamdard University (Other)
Responsible Party: Principal Investigator, Dr. Nida Shahid, Assistant Professor, Anesthesiology, Hamdard University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N0331
Record Dates: First submitted 2022-07-27; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Chills
Keywords: spinal anesthesia; vaginal hysterectomy; shivering
MeSH Terms: conditions — Chills | interventions — Dexmedetomidine; Ketamine

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to either group Dexmedetomidine (receiving I/V bolus of dexmedetomidine 0.1 mg/kg as a 20 ml solution, followed by 0.04mg/kg/hr infusion till surgery completion) OR group Ketamine (receiving 0.2 mg/kg iv of ketamine diluted to 20 ml followed by 0.1 mg/kg/hr infusion till surgery completion) through sequentially numbered opaque sealed envelope. Anesthesiologist and patients both will be blinded to the administered drug in two groups. Either of the drugs will be injected after giving spinal anesthesia and confirmation of achievement of desired level of block.
  In the recovery room Shivering grade, and vitals of patients will be evaluated every 15 minutes interval after giving the drug till 1hour postoperatively. 1st reading taken 15minutes after giving the drug will be labelled as Zero time.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: the drugs will be prepared by anesthesiologist who will not be the part of the study and these drugs will be injected by another anesthesiologist who will be blinded to the drugs and will be participating into the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Dexmedetomidine (Experimental): Group Dexmedetomidine receiving I/V bolus of dexmedetomidine 0.1 mg/kg as a 20 ml solution, followed by 0.04mg/kg/hr infusion till surgery completion
  Interventions: Drug: Dexmedetomidine
- Group Ketamine (Experimental): Group Ketamine receiving 0.2 mg/kg iv of ketamine diluted to 20 ml followed by 0.1 mg/kg/hr infusion till surgery completion
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Dexmedetomidine — I/V bolus of dexmedetomidine 0.1 mg/kg as a 20 ml solution, followed by 0.04mg/kg/hr infusion
  Arms: Group Dexmedetomidine
Drug: Ketamine — 0.2 mg/kg iv of ketamine diluted to 20 ml followed by 0.1 mg/kg/hr infusion
  Arms: Group Ketamine

SUMMARY:
comparison of Dexmedetomidine And Ketamine For Control Of Shivering In Vaginal Hysterectomy Proceeded Under Spinal Anesthesia.

DETAILED DESCRIPTION:
In this study the participants aim to Compare Dexmedetomidine And Ketamine For Control Of Shivering In Vaginal Hysterectomy Proceeded Under Spinal Anesthesia regarding efficacy, hamemodynamic stability, outcomes and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of age 45-55 years requiring vaginal hysterectomy
2. American Society of Anesthesiology (ASA) of Grade I-II

Exclusion Criteria:

1. Patients unwilling or non-cooperative for spinal anesthesia
2. Patients with uncontrolled hypertension, vascular or coronary disease,
3. patients with increased intraocular or intracranial pressure
4. Patients with known bleeding and psychiatric disorders
5. Patients taking anti platelets drugs.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female aged b/w 45-55years
Enrollment: 104 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Shivering grade | Shivering grade of patients will be evaluated every 15 minutes interval after giving the drug till 1hour postoperatively
  Shivering of patients will be grouped into five grades; Grade 0: lack of shivering, Grade I: slight shivering (inconsiderable yet apparent peripheral vasoconstriction), Grade II: medium level shivering (muscular activity in one muscle group only), Grade III: severe shivering (muscular activity in more than one muscle group without generalized shivering), Grade IV: generalized shivering.

CONTACTS AND LOCATIONS:
Overall Officials: Nida Shahid, MBBS,FCPS, Principal Investigator — Hamdard University

IPD SHARING:
Plan to Share IPD: No